CLINICAL TRIAL: NCT04555551
Title: Phase I Trial of G Protein-coupled Receptor Class C Group 5 Member D (GPRC5D) Targeted MCARH109 Chimeric Antigen Receptor (CAR) Modified T Cells for the Treatment of Multiple Myeloma
Brief Title: MCARH109 Chimeric Antigen Receptor (CAR) Modified T Cells for the Treatment of Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-367
Record Dates: First submitted 2020-09-08; First posted 2020-09-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: Adoptive T cell therapy; Chimeric Antigen Receptor; 18-367
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This phase I trial will follow a standard 3-by-3 dose escalation design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Targeted MCARH109 CAR Modified T cells (Experimental): Patients will undergo leukapheresis of peripheral blood for further T cell enrichment; activation and genetic modification using a lentiviral vector encoding a GPRC5D targeted CAR (MCARH109). These T cells will be expanded and after the appropriate number of cells is generated, the modified T cells may be infused fresh or frozen for later use according to standard operation procedures. These modified T cell infusions will be administered 2-7 days following completion of conditioning chemotherapy.
  Interventions: Biological: Infusion of MCARH109 T cells

INTERVENTIONS:
Biological: Infusion of MCARH109 T cells — Patients will be admitted to Memorial Hospital as inpatient prior to the infusion of CAR T cells. The T cell infusion will be planned to start at 2 days following the completion of the conditioning chemotherapy (up to 7 days is allowed if clinically indicated to delay).Cohorts of 3-6 patients each will be treated with escalating doses of modified T cells.

SUMMARY:
This study will test the safety of the study treatment, MCARH109, at different doses, to see which dose is safest in people, and to look for any good and bad effects of this treatment. The study treatment could stop the growth of the cancer, but it could also cause side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed MM by MSKCC pathologist.
* Age ≥ 18 years of age
* Diagnosis of relapsed or refractory multiple myeloma with at least 3 prior lines of therapy.
* Refractory myeloma is defined as disease that progresses while on therapy or within 60 days after the last therapy. Relapsed myeloma id defined as previously treated myeloma with initial response and subsequent progression (per IMWG criteria) not meeting criteria for refractory disease.
* At least 3 prior lines of therapy; Prior therapy should include all of the following-

  * A proteasome inhibitor (e.g. bortezomib, carfilzomib, ixazomib)
  * An immunomodulatory drug (e.g. thalidomide, lenalidomide, pomalidomide)
  * A CD38 monoclonal antibody (e.g. daratumumab)
  * High dose chemotherapy with autologous stem cell support (ASCT) Subjects who are not candidates to receive one or more of the above treatments are eligible for the trial
* ECOG performance status of 0 or 1
* HGB ≥ 8 g/dl, ANC≥ 1,000/mm3, Platelet≥ 50,000/mm3 without red cell transfusion for 21 days, platelet transfusion for 7 days and or growth factor support (Neupogen or Neulasta) for at least 14 days prior to initial screening (screening A). HGB ≥ 8 g/dl, ANC≥ 1,000/mm3, Platelet≥ 20,000/mm3 prior to pre-treatment screening (screening B). Patients are allowed to receive transfusion support prior to the pre-treatment screening but no growth factor support (Neupogen or Neulasta) for 7 days prior to pre-treatment screening.
* Measurable disease defined as meeting at least one of the criteria below-

  * Serum M protein ≥ 0.5 g/dL
  * Involved serum free light chain ≥10 mg/dL with an abnormal free light chain ratio
  * Urine M-protein ≥ 200 mg/24 hours
  * Measurable plasmacytomas seen on imaging (≥ 1 lesion that has a single diameter ≥ 2 cm) If this is the primary marker of measurable disease, patients will need a biopsy at the pre-treatment screening (screening B).
  * Bone marrow plasma cells ≥ 30% as determined by CD138 immunohistochemistry staining
* Serum creatinine ≤ 1.5mg/dL or a measured creatinine clearance ≥ 50 mL/min (using 24-hour urine collection)
* ALT and AST ≤ 3 X ULN and total bilirubin ≤ 2 mg/dL (or < 3 mg/dL for individuals with Gilbert's syndrome)
* PT and PTT ≤ 1.5 X ULN
* Adequate pulmonary function as assessed by ≥92% oxygen saturation on room air by pulse oximetry
* Adequate cardiac function, defined as LVEF ≥ 40% by echocardiogram performed within 4 weeks of initial screening
* For patients with prior ASCT, at least 100 days since ASCT at the time of initial screening

Exclusion Criteria:

* Pregnant or lactating women. Women and men of childbearing age should use highly effective contraception while on this study and continue for 1 year after all treatment is finished.
* Patients with following cardiac conditions will be excluded:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure
  * Myocardial infarction ≤6 months prior to enrollment
  * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
  * History of severe non-ischemic cardiomyopathy
* Patients with HIV or active hepatitis B or hepatitis C infection are ineligible.
* Current diagnosis of primary and secondary plasma cell leukemia is excluded. History of plasma cell leukemia is not excluded.
* Patients who have not received any myeloma therapy for the preceding 6 months, except if the last myeloma therapy was a CAR T cell therapy.
* At least 14 day washout from myeloma therapies prior to leukapheresis and prior to starting lymphodepletion. The washout for experimental treatments would be 5 half lives or 14 days (whichever is shorter).
* At least 14 day washout from radiation prior to leukapheresis and prior to starting lymphodepletion.
* Patients treated with previous GPRC5D targeted therapies would be excluded.
* Patients with any concurrent active malignancies (or another primary malignancy not in remission for at least 2 years) as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of skin.
* Patients with a prior allogeneic transplant at least 6 months prior to study enrollment ARE eligible UNLESS experienced GvHD that required systemic steroids or other systemic lymphotoxic therapy within 12 weeks of initial screening
* Patients on systemic steroids (except if solely for adrenal replacement) within two weeks of collection
* Active auto-immune disease including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis, or have a history of severe (as judged by the principal investigator) autoimmune disease requiring prolonged immunosuppressive therapy
* Prior or active CNS involvement by myeloma (e.g. leptomeningeal disease). Screening for this, for example, by lumbar puncture, is only required if suspicious symptoms or radiographic findings are present.
* Pre-existing (active or severe) neurologic disorders (e.g. pre-existing seizure disorder)
* Active uncontrolled acute infections
* Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 1 year
  The MTD is defined as the highest dose with an observed incidence of DLT in no more than one out of six patients treated at a particular dose level. All patients treated in a dose cohort will be observed a minimum of 30 days before the T cell dose can be escalated.

SECONDARY OUTCOMES:
overall response rate (ORR) | approximately 1 and 4 weeks following the T cell infusion
  Assessed by the IMWG 2016 criteria.The major criteria for determination of response to therapy in patients with MM include examination of the peripheral blood and bone marrow. Bone marrow aspirate and biopsy obtained at approximately 1 and 4 weeks following the T cell infusion will be used for disease response assessment. Definitions for response assessment will be as defined by the pending update to the international myeloma working group (IMWG) guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Sham Mailankody, MBBS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Jurgens EM, Firestone RS, Chaudhari J, Hosszu K, Devlin SM, Shah UA, Landa J, McAvoy DP, Lesokhin AM, Korde N, Hassoun H, Tan CR, Hultcrantz M, Shah GL, Landau HJ, Chung DJ, Scordo M, Eren OC, Dogan A, Giralt SA, Park JH, Riviere I, Brentjens RJ, Smith EL, Wang X, Usmani SZ, Mailankody S. Phase I Trial of MCARH109, a G Protein-Coupled Receptor Class C Group 5 Member D (GPRC5D)-Targeted Chimeric Antigen Receptor T-Cell Therapy for Multiple Myeloma: An Updated Analysis. J Clin Oncol. 2025 Feb 10;43(5):498-504. doi: 10.1200/JCO-24-01785. Epub 2024 Dec 4. PMID 39631041
- [Derived] Mailankody S, Devlin SM, Landa J, Nath K, Diamonte C, Carstens EJ, Russo D, Auclair R, Fitzgerald L, Cadzin B, Wang X, Sikder D, Senechal B, Bermudez VP, Purdon TJ, Hosszu K, McAvoy DP, Farzana T, Mead E, Wilcox JA, Santomasso BD, Shah GL, Shah UA, Korde N, Lesokhin A, Tan CR, Hultcrantz M, Hassoun H, Roshal M, Sen F, Dogan A, Landgren O, Giralt SA, Park JH, Usmani SZ, Riviere I, Brentjens RJ, Smith EL. GPRC5D-Targeted CAR T Cells for Myeloma. N Engl J Med. 2022 Sep 29;387(13):1196-1206. doi: 10.1056/NEJMoa2209900. PMID 36170501
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm